CLINICAL TRIAL: NCT04932135
Title: Resting Heart Rate Monitoring for Optimized Treatment and Surveillance of Hyperthyroidism
Acronym: PULSAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2021-00422
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hyperthyroidism; Graves Disease
Keywords: Heart rate; Pulse rate
MeSH Terms: conditions — Hyperthyroidism; Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Treatment: Patients with newly diagnosed hyperthyroidism due to Graves' disease, if anti thyroid drug treatment is planned.
  Interventions: Diagnostic Test: Continuous heart rate monitoring
- Group Surveillance: Patients suffering from Graves' disease in whom discontinuation of the anti-thyroid therapy is planned.
  Interventions: Diagnostic Test: Continuous heart rate monitoring

INTERVENTIONS:
Diagnostic Test: Continuous heart rate monitoring — Continuous heart rate monitoring with a wrist worn fitnesstracker
  Other Names: Regular measurements of thyroid hormone levels

SUMMARY:
The investigators want to investigate if a continuous heart rate monitoring with a wrist worn fitnesstracker can be useful in the treatment and surveillance of patients suffering from Graves' disease.The aim of our research project is two-fold: First, to evaluate the use of continuous heart rate monitoring as a potential substitute for hormone measurements during treatment of hyperthyroidism. Second, to use continuous heart rate monitoring as a tool for early detection of relapse after discontinuation of antithyroid drugs.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* BMI 17 to 35 kg/m2
* Diagnosis of Graves' disease (matching one of the following criteria: elevated TRAb and/or ultrasonography and functional imaging consistent with Graves' disease)
* In possession of a smart phone
* Able to use a wearable device and willing to regularly upload their biometric data
* Informed consent as documented by signature (Appendix Informed Consent Form)

Group "treatment":

* TSH < 0.2 mIU/l and
* fT4 > 25 pM or fT3 > 8 pM
* ATD planned, additional treatment with propranolol allowed

Group "surveillance":

* TSH within the reference range between 0.3 and 4.5 mlU/l
* Cessation of ATD is planned within the next 2-4 weeks

Exclusion Criteria:

* Chronic treatment with beta blocker or verapamil-type calcium antagonist for other reason than symptomatic treatment of hyperthyroidism (propranolol)
* Treatment with amiodarone
* Pacemaker with continuous stimulation.
* Severe concomitant diseases: chronic heart failure, liver cirrhosis, kidney failure, active cancer
* Abuse of alcohol or illicit drugs
* Allergic to nickel or silicone
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Graves' disease at the beginning and after cessation of anti-thyroid drug treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
resting heart rate | four months
  continuous resting heart rate measurement with fitnesstracker in relation to the thyroid hormone levels in patients during and after treatment with anti-thyroid drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No